CLINICAL TRIAL: NCT04384809
Title: Comparison of Leukocyte-rich Platelet Rich Plasma Injection to Percutaneous Tenotomy in the Treatment of Chronic Common Extensor Tendinopathy
Brief Title: Platelet Rich Plasma Injection vs Percutaneous Tenotomy for Common Extensor Tendinopathy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20200165
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: common extensor; lateral epicondyle; tennis elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Non-blinded, parallel randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Leukocyte rich platelet rich plasma injection (Experimental): Patients will be injected with leukocyte rich platelet rich plasma in their common extensor tendon
  Interventions: Biological: Leukocyte rich platelet rich plasma
- Percutaneous tenotomy (Experimental): Patients will undergo percutaneous tenotomy of the common extensor tendon using the Tenex tenotomy device
  Interventions: Device: Percutaneous Tenotomy

INTERVENTIONS:
Biological: Leukocyte rich platelet rich plasma — Leukocyte rich platelet rich plasma will be obtained and prepared from a peripheral artery of the subject and then will be injected in the common extensor tendon
  Arms: Leukocyte rich platelet rich plasma injection
Device: Percutaneous Tenotomy — Patients will undergo percutaneous tenotomy of the common extensor tendon using the Tenex tenotomy device
  Arms: Percutaneous tenotomy

SUMMARY:
This is a randomized control trial comparing the use of leukocyte rich platelet rich plasma injections to percutaneous tenotomy for the treatment of chronic common extensor tendinopathy.

DETAILED DESCRIPTION:
This is a randomized control trial comparing the use of leukocyte rich platelet rich plasma injections to percutaneous tenotomy for the treatment of chronic common extensor tendinopathy. Patients with a history of common extensor tendinopathy for greater than 3 months, refractory to conservative treatments, are randomized into one of two groups: injection with leukocyte rich platelet rich plasma or percutaneous tenotomy with the Tenex system. Both groups of patients are followed up in clinic at 1 week, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year following the procedure to examine levels of pain or complications following both procedures.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of lateral elbow pain
* Subjectively failed trial of physical therapy and counterbracing
* Identifiable pathology on ultrasound (one or more of the following: thickened or disorganized tendon origin, microtearing, edema, neovascularization

Exclusion Criteria:

* Steroid injection within the last 3 months
* Previous surgery for common extensor tendinopathy
* Current treatment with analgesics
* Pregnant, non-English speaking, or illiterate individuals
* History of anemia
* History of bleeding disorder
* Anticoagulant use
* History of cervical radiculopathy
* Hemoglobin less than 11 grams per deciliter
* Hematocrit less than 33%
* Platelet count outside of normal range of 150-400 x 1000 microliter

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain: visual analogue scale | up to 12 months post-procedure
  Change in pain will be measured using a 10 point visual analogue scale where 0 represents no pain and 10 indicates the worst pain possible.
Change in function | up to 12 months post-procedure
  Change in function will be measured using the Oxford Elbow score using a 48 point scale where a score of 0 indicates severe functional impairment and a score of 48 indicates no functional impairment

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States